CLINICAL TRIAL: NCT00005637
Title: A Phase I Study of Extended Low Dose Temozolomide (SCH 52365, Temodar (R)) and Carmustine (BCNU) in the Treatment of Malignant Gliomas After Radiation Therapy
Brief Title: Combination Chemotherapy Following Radiation Therapy in Treating Patients With Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067793; MSKCC-99114; NCI-G00-1765
Record Dates: First submitted 2000-05-02; First posted 2003-01-27 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2003-03

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult giant cell glioblastoma; adult gliosarcoma; adult anaplastic ependymoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma; Gliosarcoma; Ependymoma | interventions — Carmustine; Temozolomide

INTERVENTIONS:
Drug: carmustine
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one chemotherapy drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy following radiation therapy in treating patients who have malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and efficacy of extended low-dose temozolomide when combined with carmustine after radiotherapy in patients with malignant glioma.
* Determine the maximum tolerated dose of this combination in this patient population.
* Determine time to progression as measured from baseline gadolinium-enhanced magnetic resonance imaging in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of temozolomide.

Patients receive oral temozolomide once daily on days 1-28 and carmustine IV over 1-3 hours beginning within 72 hours after starting temozolomide. Courses repeat every 8 weeks for up to 1 year in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating doses of temozolomide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 3-24 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant glioma

  * Glioblastoma
  * Gliosarcoma
  * High-grade glioma
  * Anaplastic astrocytoma
  * Anaplastic mixed oligoastrocytoma
  * Anaplastic oligodendroglioma
  * Anaplastic ependymoma
* Must have completed radiotherapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* More than 3 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* SGOT/SGPT less than 3 times ULN
* Alkaline phosphatase less than 2 times ULN

Renal:

* BUN less than 1.5 times ULN
* Creatinine less than 1.5 times ULN

Pulmonary:

* Pulmonary function test with diffusion greater than 50 OR
* Clearance by the pulmonary service

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No AIDS-related illness
* No nonmalignant systemic disease that would preclude study
* No acute infection requiring IV antibiotics
* No psychiatric condition that would preclude study compliance
* No frequent vomiting or medical condition that would interfere with oral medication intake (e.g., partial bowel obstruction)
* No other prior or concurrent malignancy except surgically cured carcinoma in situ of the cervix or basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy
* No prior biologic therapy

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 2 weeks since prior radiotherapy

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-12; Primary Completion 2003-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J. Raizer, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States